CLINICAL TRIAL: NCT02912637
Title: Hyperpolarised 129Xe MRI for Non-invasive Assessment of Ventilation, Perfusion and the Alveolar Membrane - a Physiological Study in Healthy Volunteers & Cystic Fibrosis Patients
Brief Title: Hyperpolarized Xenon Imaging in Patients With Cystic Fibrosis
Status: Withdrawn | Type: Observational
Why Stopped: Technical and administrative problems
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: P02215
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- CF patients: Hyperpolarized Xenon MRI
  Interventions: Other: Hyperpolarized Xenon MRI
- Healthy volunteers: Hyperpolarized Xenon MRI
  Interventions: Other: Hyperpolarized Xenon MRI

INTERVENTIONS:
Other: Hyperpolarized Xenon MRI — MRI & MRS of lung using inhaled hyperpolarized Xenon as a contrast agent

SUMMARY:
Chronic lung diseases show a gradual onset of irreversible lung damage which can lead to severe breathing problems and/or respiratory failure. Imaging is central to guiding treatment; however, current techniques are either inaccurate or involve exposure to radiation. Recent developments in lung magnetic resonance imaging (MRI) provide promise as a radiation-free alternative. However, conventional MRI cannot directly show changes in distribution of inhaled air or absorption of gas which are important signs of early lung disease. Recently MRI imaging of the inhaled gas contrast agent Xenon has been developed which can provide this important information. This study aims to determine how Xenon MRI can help determine air flow distribution and gas uptake in the lungs. The investigators will also be able to compare the information from patients with that from healthy volunteers. This should give insight into the processes involved in chronic lung diseases and help evaluate disease extent in patients.

DETAILED DESCRIPTION:
Hyperpolarised gas MRI (3He and 129Xe) has enabled novel methods of in-vivo functional lung imaging that do not rely on the use of ionising radiation. Hyperpolarised 129Xe (HP Xe) MRI provides additional complementary information to 3He and 1H MRI and conventional lung imaging modalities. By virtue of its solubility, the 129Xe contrast agent follows the gas exchange pathways in the lungs, offering a direct means to explore regional ventilation-perfusion (V/Q). The competing modality of nuclear medicine lung V/Q scans suffer from very poor spatial resolution and a reliance on high doses of radiation via radio-nuclide inhalation. Nuclear medicine is thus unsuitable for studies of basic physiology in healthy volunteers or in longitudinal studies in lung disease patients.

The aims and objectives of this study are:

1. To assess the physiological differences in lung ventilation between the normal group (volunteers) and the cystic fibrosis disease group
2. To evaluate differences in Xe diffusion across the alveolar membrane between the normal group (volunteers) and the cystic fibrosis disease group
3. To understand the relationship between the extent of abnormal ventilation (and ventilation-perfusion mismatch) on MRI and the results from conventional physiological evaluation of lung function using pulmonary function tests (spirometry and gas exchange)
4. To understand the relationship between gas exchange as determined by HP Xe imaging with the extent of ventilation perfusion mismatch on standard perfusion MRI

This is a physiological cross-sectional feasibility study comparing regional lung ventilation and diffusion across the alveolar membrane in normal volunteers and cystic fibrosis. 15 healthy volunteers and 15 cystic fibrosis patients will be recruited. All imaging will take place at Papworth Hospital.

Phase I: Volunteer study (n=15, aged 18-70)

Hyperpolarised 129Xe MRI scans will be performed in the MRI department at Papworth Hospital, using a Siemens Avanto 1.5 Tesla system with 129Xe capability using a dedicated transmit-receive RF coil.

Phase II: CF study (n=15, aged 18-70)

Patients already enrolled in the study 'Pulmonary magnetic resonance imaging in cystic fibrosis: accuracy and reproducibility' (REC reference: 13/EE/0401; IRAS project ID: 73137) will be invited to take part in this study too.

These patients, with CF in stable phase, will be evaluated with same day conventional MRI, lung function tests and clinical scoring. The methodology of 129Xe MRI will be as described above for healthy volunteers.

Morphological imaging: A combination of T1 and T2 weighted sequences will be used.

Hyperpolarized 129Xe MR imaging: For each subject, up to two deliveries of ≤ 1L doses of hyperpolarised xenon will take place as follows:-

1. 129Xe ventilation imaging will provide further information on assessment of lung ventilation volume using a volumetric gradient echo sequence.
2. Chemical shift saturation recovery (CSSR) spectroscopy with dissolved xenon will provide an estimation of the fraction of 129Xe in tissue/interstitium and in red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above with proven CF, and:
* Clinical stable disease over last month, defined as:

One month without intravenous antibiotics for airways disease, and:

One month without evidence for decrease in lung function (no evidenced drop in FEV1 or PEFR >10%).

Exclusion criteria:

* Contraindications to MR (presence of non MR compatible pacemaker, aneurysm clips, artificial heart valves, ear implants, metal fragments or metallic foreign objects in the eyes, pregnancy, and severe claustrophobia),
* Ability to breath hold below 15 seconds.
* Current (> 6 months) smoker

Volunteer inclusion criteria:

* No history of acute (within the last 6 months) or chronic illness (this will be determined by direct communication with the volunteer and not from their medical records)

Volunteer exclusion Criteria:

* As patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cystic fibrosis and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Lung ventilation assessed by Percentage Ventilation Defect (VD%) | 24 hours
  Quantitative measure of lung ventilation

SECONDARY OUTCOMES:
Forced expiratory volume (%) in 1 second (FEV1) | 24 hours
  Quantitative measure of lung function
Percentage perfusion defect (PD%) | 24 hours
  Quantitative measure of lung perfusion
Regional ventilation: perfusion (1-VD%)/(1-PD%) ratio | 24 hours
  Quantitative measure of regional lung function
CF Brody score assessed on CT in patient group | 24 hours
  Disease severity (in patients) assessed by routine CT
Percentage ventilation defect assessed on CT (hypoattenuation) - patient group only | 24 hours
  Disease severity (in patients) assessed by quantitative measure of ventilation on routine CT

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Screaton, Principal Investigator — Papworth NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No